CLINICAL TRIAL: NCT03421223
Title: Digital Signals in Chronic Pain (DiSCover Project)
Status: Completed | Type: Observational
Sponsor: Evidation Health (Industry)
Responsible Party: Sponsor
Other Study IDs: EH-007
Record Dates: First submitted 2018-01-07; First posted 2018-02-05 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Individuals diagnosed with chronic pain
  Interventions: Other: No intervention
- Control: Individuals without chronic pain
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The DiSCover Project is a 1-year longitudinal case-control observational study. In this study, the investigators plan to collect different types of data including self-reported health outcomes and quality of life data, behavioral data from activity trackers and health and fitness apps, data from lab tests, genetic data, and environmental data. One of the goals of this study is to develop digital biomarkers for chronic pain severity, flare ups and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Resides in the United States
* Case Inclusion Criteria: Self-reported diagnosis of chronic pain and experiences moderate chronic pain as assessed by scoring at least 4 on the Numeric Pain Rating Scale
* Control Inclusion Criteria: Self-reported not having chronic pain

Exclusion Criteria:

* Less than 18 years old
* Is not able to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit virtually and individuals can participate remotely.
Sampling Method: Non-Probability Sample
Enrollment: 10161 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Self-reported chronic pain severity measured by BPI-SF | 1 year
Quality of Life Scale for Pain | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jessie L Juusola, PhD, Principal Investigator — Evidation Health
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No